CLINICAL TRIAL: NCT01161719
Title: The Effectiveness of Videoconferencing on Teaching Parent Training Skills to Parents of Children With ADHD
Brief Title: Effectiveness Study of Videoconferencing on Teaching Parent Training Skills to Parents of Children With Attention Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200816003
Record Dates: First submitted 2010-06-25; First posted 2010-07-13 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; Parent training; Videoconference
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Videoconference (Experimental): Parent training through videoconference
  Interventions: Behavioral: parent training
- Control (Active Comparator): Parent training through face to face conference
  Interventions: Behavioral: parent training

INTERVENTIONS:
Behavioral: parent training — Behavioral management skill training

SUMMARY:
The purpose of this study is to evaluate the effectiveness of group parent training taught through videoconferencing on ADHD treatment via a comparison between participants using traditional face-to-face parent training sessions and a group using teleconferencing.

DETAILED DESCRIPTION:
Subjects with a primary diagnosis of ADHD between the ages of 6 and 14 years were enrolled. All subjects were screened and assessed for psychiatric and learning disorders using structured interviews (DICA, parent and child version, Reich et al, 2000) based on DSM IV criteria and parent and teacher rating scales. Mothers took the Beck Depression Inventory (BDI) to assess for depression.

Parents or primary caregivers were randomized to two treatment arms (videoconference or face to face). Ten sessions of weekly parent training through either videoconference or face-to-face delivery was conducted using Dr. Russell A. Barkley's manual. A non-mandatory skill training and play group was offered to the children of both groups while parents attended the parent training group in order to provide child care for the parents during the training sessions.

Following outcomes will be measured to assess the effectiveness of the intervention:

Primary outcome Acceptance of the parent and children on the mode the communication as well as parent training.

Secondary outcomes:

1. Parent-child relations measured by the Parent Child Relationship Questionnaire (PCQ)
2. The Vanderbilt Assessment Scale (parent & teacher versions), Children Global Assessment Scale (CGAS), Clinical Global Impression- Severity score (CGI-S), and Clinical Global Impression-Improvement Scores (CGI-I) assessed the severity of core symptoms of ADHD and oppositional/aggressive symptoms.
3. The parent and teacher-rated versions of the Social Skills Rating System (SSRS) assessed social skills.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV criteria for any subtype of ADHD.
* ADHD must be the primary diagnosis if there is comorbidity.

Exclusion Criteria:

* Subjects with significant medical conditions, which are not stable on current outpatient treatment regimen.
* Subjects with severe psychiatric disorders (i.e., bipolar disorder, autism, schizophrenia, major depression).

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2008-04; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Acceptance of the parent and children on the mode the communication as well as parent training | One year
  Acceptance of the parent and children on the mode the communication as well as parent training will be measured by a Likert scale, which is a 12 intem questionaire to assess parent's satisfaction with the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Yuhuan Xie, MD, Principal Investigator — University of California, Davis
Locations (1):
- UC Davis MIND Institute, Sacramento, California, United States

REFERENCES:
- [Derived] Xie Y, Dixon JF, Yee OM, Zhang J, Chen YA, Deangelo S, Yellowlees P, Hendren R, Schweitzer JB. A study on the effectiveness of videoconferencing on teaching parent training skills to parents of children with ADHD. Telemed J E Health. 2013 Mar;19(3):192-9. doi: 10.1089/tmj.2012.0108. Epub 2013 Feb 13. PMID 23405952